CLINICAL TRIAL: NCT05706142
Title: Motor Imagery on Learning Infant Massage
Brief Title: Determination of the Effects of Motor Imagery on Learning Infant Massage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ETK00-2022-0275
Record Dates: First submitted 2023-01-11; First posted 2023-01-31 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Students
Keywords: physiotherapy and rehabilitation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): No motor imagery will be shown to these students. The same massage will only be shown as practically at class.
- Intervention Group (Experimental): Within the scope of motor imagery training, a presentation will be made to the students of pediatric rehabilitation lecture in the intervention group about what motor imagery is. "PETTLEP" model will be used for imagery training. In this model, imagery training will be prepared in accordance with our purpose, taking into account the physical, environmental, time, task, learning, emotion and personal subheadings. In the training sessions, relaxation exercises will be given for 5 minutes first. After the relaxation exercises, special "colic massage" imagery training will be given to newborns for 10 minutes. The massage will also be shown as practically at class.
  Interventions: Other: Motor Imagery Education

INTERVENTIONS:
Other: Motor Imagery Education — Within the scope of motor imagery training, a presentation will be made to the students of pediatric rehabilitation lecture in the intervention group about what motor imagery is. "PETTLEP" model will be used for imagery training. In this model, imagery training will be prepared in accordance with our purpose, taking into account the physical, environmental, time, task, learning, emotion and personal subheadings. In the training sessions, relaxation exercises will be given for 5 minutes first. After the relaxation exercises, special "colic massage" imagery training will be given to newborns for 10 minutes. The massage will also be shown as practically at class.
  Arms: Intervention Group

SUMMARY:
Motor imagery is the mental rehearsal of simple or complex motor movements in which no clear body movement occurs. It can also be defined as the mental simulation of movement without revealing any real motor movement. Studies have shown that similar brain regions are activated during the performance of the movement and the imagery of the movement. According to the results obtained from advanced imaging techniques, it has been reported that activations occur in similar areas during motor imagery and physical performance, including brain areas such as premotor areas, parietal lobe, basal ganglia, anterior cingulate cortex, and cerebellum. When the literature is examined, it has been seen that motor imagery applications are used in many different areas. In 2021, the effect of motor imagery training on students' motor imagery levels and practice in the education of medical school students by Collet et al. was investigated. As a result of the training, it was reported that motor skills improved and it strengthened the learning of medical skills.

DETAILED DESCRIPTION:
Infantile colic was first defined in 1954 by Wessel et al. The incidence of infantile colic varies between 10-30%. There was no study showing the general colic frequency in Turkey, however, in a study conducted in the Eastern Anatolia Region in 2005, the incidence of infantile colic was reported as 51.1%. Although the causes of colic are not fully explained, food allergy or lactose intolerance, hypersensitivity, abnormal peristalsis or excessive gas, tension and stress in the family, swallowing air during bottle feeding or excessive crying, gastro-esophageal reflux, low birth weight, psychosocial It is thought that factors such as problems cause colic.

Thus, in physiotherapy education, there are many practical lectures. In the recent years, motor imagery has been used to teach exercises to the patients who need physiotherapy like stroke patients. Thus, it is considered that motor imagery can be used in the education and in the literature, there are papers which investigate the effects of motor imagery among the students of nursing and medicine. In conclusion, the aim is to see whether this method can be used as a new teaching method among physiotherapy students, thus this may bring the students more familiar for the use in their future clinical practices.

ELIGIBILITY:
Inclusion Criteria:

* Individuals over the age of 18
* To be taking the Pediatric Rehabilitation course for the first time in the Fall semester of the academic year 2022-2023 at the Eastern Mediterranean University, Department of Physiotherapy and Rehabilitation.

Exclusion Criteria:

* Having serious vision and hearing problems,
* Having serious attention problems,
* Having a musculoskeletal, cardiovascular, pulmonary, metabolic, or other disease severe enough to preclude participation in the study.
* Prior participation in any kind of motor imagery training

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Motion Imagery Questionnaire | change from baseline at two weeks study duration
  The Motion Imagery Questionnaire-3 is an adaptation of the Motion Imagery Questionnaire. It consists of 3 subscales and a total of 12 items evaluating external visual imagery, internal visual imagery and kinesthetic imagery. Before starting the evaluation, the participants are given the necessary information about the survey. Each of the 12 tasks in the questionnaire is performed physically first, then the participant returns to the starting position and visualization is performed according to the desired imagery type. The scoring is between 1 and 7, with 1 point: very difficult to see/feel, 7 points: very easy to see/feel. While calculating the score, the internal visual imagery, external visual imagery and kinesthetic imagery scores are added separately and divided by 4 and averaged. Higher scores show better imagery ability.

SECONDARY OUTCOMES:
Chronometry for colic massage on baby doll | change from baseline at two weeks study duration
  Individuals participating in the study are asked to perform colic massage actively on baby dolls. They are asked to record this time in seconds.
Mental Chronometry for colic massage | change from baseline at two weeks study duration
  They are asked to visualize the colic massage using internal and then external perspective. The time visualised is recorded in seconds.
Proportion between real and mental chronometry | change from baseline at two weeks study duration
  The proportion is taken between the real massage and imagined massage.
Qualitative effects | at two weeks
  The students in the intervention group will be asked to reply five open ended questions about the effects of motor imagery on learning colic massage for infants. The Microsoft Teams will be used for voice record with the feature of "speech to test".

CONTACTS AND LOCATIONS:
Overall Officials: Zehra Güçhan Topcu, Assist.Prof., Principal Investigator — Lecturer at university
Locations (2):
- Eastern Mediterranean University, Famagusta, Güney Kampüs, Cyprus
- Eastern Mediterranean University, Faculty of Health Sciences, Physiotherapy and Rehabilitation Department, Mersin, Famagusta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No